CLINICAL TRIAL: NCT05072834
Title: Identification of Novel Biomarkers for Environmental Enteropathy in Children Using an Evidence Based Approach
Brief Title: Identification of Novel Bio-markers for Environmental Enteropathy in Children Using an Evidence Based Approach
Acronym: EE
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Collaborators: University of Reading (Other); Boston University (Other); Washington University School of Medicine (Other); University of Chicago (Other); University of Virginia (Other)
Responsible Party: Principal Investigator, Dr Syed Asad Ali, Assistant Professor, Aga Khan University
Other Study IDs: 12-2012
Record Dates: First submitted 2015-06-26; First posted 2021-10-11 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Malnutrition; Enteropathy
Keywords: Environmental Enteropathy; Childhood malnutrition; biomarkers
MeSH Terms: conditions — Malnutrition; Intestinal Diseases | interventions — Endoscopy, Digestive System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — collect blood, urine and stools at 6 and 9 months of age and test for biomarkers including GLP-2, Claudin 3, CRP, Reg 1, serum cytokines profile, plasma amino acids profile, Neopterin and Myeloperoxidase
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cohort A: children with chronic malnutrition who do not respond to adequate supplemental feeding will undergo Upper Gastrointestinal Endoscopy
  Interventions: Procedure: Upper Gastrointestinal Endoscopy
- Cohort B: Children 6 months to 24 months old who are undergoing Upper Gastrointestinal endoscopy for any appropriate indication
  Interventions: Procedure: Upper Gastrointestinal Endoscopy

INTERVENTIONS:
Procedure: Upper Gastrointestinal Endoscopy — Procedure Upper gastro-intestinal endoscopic procedure involves collection of intestinal samples and it can be helpful in identifying the causes of malnutrition. Upon parental approval, the child along with two relatives will be provided transportation to Karachi, accommodation and the compensation for their time and expenses.
  For this procedure the child will be admitted to the hospital a day before the procedure till one day after the procedure. This procedure takes 30 minutes, requires general anesthesia and involves insertion of a flexible tube with a small TV camera and a light on one end and an eyepiece on the other. The endoscope will allow the doctor to examine the inside of certain tube-like structures in the body. Some tissue samples for laboratory testing will be taken.
  Other Names: UGI endoscopy

SUMMARY:
EE is increasingly recognized as a key factor underlying malnutrition, weakened immune response and impaired cognitive development in children in developing countries. Absence of a distinct biomarker of EE in the blood, urine or stool makes it difficult to study the impact of interventions against it. Biomarkers for EE have been challenging to find, partly because of our inadequate understanding of its pathophysiology. Investigators aim to identify novel biomarkers for EE, based on our hypothesis that EE is a result of two processes: 1) repeated exposure to enteric pathogens and environmental toxins leading to gut inflammation and 2) weaning on diets high in carbohydrates but low in proteins and fat, leading to atrophy of the intestinal mucosa. This leads to gut dysfunction, including leaky gut, small bowel stasis, bacterial overgrowth, decreased immune response to infections, and frequent diarrhea. The candidate biomarkers investigators have selected for our study (CRP, GLP- 2, Claudin 3, Reg-1, plasma amino acids profile, serum cytokine profile, Neopterin and Myeloperoxidase) are markers of inflammation, hormonal dysfunction and tight junction malfunction of the small intestines. The 'gold standard test' for EE will be direct histopathologic analysis of the duodenal mucosa, which will be available in a subset of study children undergoing upper GI endoscopy. For other study subjects, clinical surrogates for EE will be used to calculate the sensitivity and specificity of biomarkers being tested. These clinical surrogates of EE include HAZ and WAZ score < 2 SD at 12 months and 15 months of age, and the worsening in HAZ and WAZ scores between 6, 9, 12 and 15 months of age. Investigators plan to study and compare duodenal biopsies from children with and without EE using cutting edge technologies including electron microscopy, immunofluorescence, and mRNA sequencing. This will allow direct correlation of the biomarkers in the blood, urine and stools with the histopathologic features of the gut mucosa. The mRNA sequencing of the gut tissue will allow us to identify new evidence-based biomarkers for EE, which could be further tested in the future.

This is a strong, multidisciplinary collaboration between investigators in Pakistan and the United States with expertise in complementary areas including chemokines, inflammation, gut architecture, infectious diseases, field studies, and technology development.

DETAILED DESCRIPTION:
Title of protocol:

Identification of Novel Biomarkers for Environmental Enteropathy in Children using an Evidence Based Approach

Background

Childhood malnutrition is a major problem in third world countries. One of the primary mechanisms behind childhood malnutrition is that consumption of low quality food and frequent gastrointestinal (GI) infections damage the intestinal mucosa of children. The intestines are thus not able to absorb the available nutrients and also fail to function as an effective barrier against the translocation of GI flora into the systemic circulation. The limited energy resources available to the child are diverted to overcome these inflammatory challenges at the expense of normal growth. This disorder of intestines (enteropathy) is called Environmental Enteropathy (EE). Since EE is thought to be a precursor of chronic malnutrition, detecting EE early with the use of biomarkers in the blood, urine or stools will allow us to predict chronic malnutrition in children early. The purpose of this research is to identify biomarkers for EE.

Objectives

1. To test novel candidate biomarkers of EE in a cohort of children 6-15 months of age in a rural district in Pakistan.
2. To study the histo-pathologic characteristics of small bowel mucosa of moderate to severely malnourished children of the study cohort A, and correlate findings with the biomarkers studied in aim 1.
3. To study the histo-pathologic characteristics of small bowel mucosa of children (well-nourished or malnourished) who are undergoing UGI endoscopy for any clinical indication e.g. retrieval of foreign body, evaluation of UGI bleeding etc., (cohort B) and correlate the findings with the blood, urine and stool biomarkers studied in aim 1.
4. To identify new candidate biomarkers for EE through studying mRNA expression in the small bowel mucosa of children with and without EE for wide range of proteins involved in inflammation, hormonal dysfunction, immune system and tight junction structure and function.

Methods

In a cohort of children already being followed for growth and infections since birth for the RESPAK study in Matiari, Sindh (Cohort A), investigators will collect blood, urine and stools at 6 and 9 months of age and test for biomarkers including GLP-2, Claudin 3, CRP, Reg 1, serum cytokines profile, plasma amino acids profile, Neopterin and Myeloperoxidase. These biomarkers will be correlated with clinical surrogates of EE, including Height for Age Z score (HAZ) and Weight for Age Z score (WAZ) of children at 6, 9, 12 and 15 months of age, and the change in HAZ and WAZ scores between 6, 9, 12 and 15 months of age Investigators will identify 20-30 children within cohort A who are moderately or severely malnourished and have history of frequent or prolonged diarrhea at 10 -11 months of age, whose diagnosis remains unknown despite a comprehensive non-invasive workup and who fail to respond to first line of nutritional interventions. These children will undergo upper GI endoscopy at the Aga Khan University, in line with the American Society for Gastroenterologlists (ASGE) guidelines for the evaluation of children who are FTT and have associated frequent or prolonged diarrhea(1). The duodenal biopsies obtained through the endoscopies will be used for H&E staining (standard of care to diagnose celiac disease, other inflammatory and autoimmune causes of enteropathy) as well as EE research, including study of inflammation, hormone dysfunction and tight junction malfunction at AKU, University of Chicago and University of Virginia.

In a separate cohort of children (Cohort B) 6-24 months old who present to our collaborating pediatric gastroenterologists at the Aga Khan University or at Children's Hospital Lahore for UGI endoscopy for any appropriate indication, additional duodenal biopsies and blood/urine/stool samples will be collected after informed consent. The workup done on these children will be as described above.

The RNA will be extracted from the entire biopsy specimen obtained, and the mRNA targets which are differentially expressed in children with and without EE will be identified, so their downstream proteins could be identified and tested as candidate biomarkers for EE in the future.

Adverse effects

Obtaining blood, urine and stools from the child at 6 and 9 months of age will cause discomfort to the child though any serious adverse event resulting from these procedures is unlikely. For subjects not responding to nutritional rehabilitation, and in whom the first line of diagnostic workup is unrevealing, advanced workup will be offered per the ASGE guidelines, which include UGI endoscopy in selected cases. Although rare, risks of endoscopy include general anaesthesia related complications, perforation, bleeding and infection.

Ethical issues

Besides the issue of privacy invasion and blood, urine and stool collection, the major ethical challenge in cohort A is the conduct of UGI endoscopies in some children in whom cause of malnutrition is unclear despite first line of investigations and interventions. Investigators think that these endoscopies are in the interest of these children, since the ASGE recommends them as part of the workup in children who are failing to thrive and have gastrointestinal symptoms like chronic or recurrent diarrhoea. The endoscopies may help identify treatable inflammatory, infectious or autoimmune causes of failure to thrive in these children.

Investigators are collecting additional biopsies for research during the endoscopies. The risks associated with endoscopy are primarily with anaesthesia and procedure. Taking additional biopsies is relatively safe since GI mucosa is one of the fastest healing organs of the body and essentially no residual sign of the biopsy is left after 24 hours of the procedure. Endoscopies at AKU and Children's hospital will be conducted by expert paediatric gastroenterologists. Nonetheless, investigators are well equipped to handle any complication that may arise.

In cohort B, investigators are taking additional biopsies from children who are already undergoing UGI endoscopies for an appropriate indication not related to this study. The only additional risk to the subjects in cohort B is with taking additional biopsies, which should be minimal as explained above.

ELIGIBILITY:
Inclusion Criteria:

1. chronically malnourished children at 9 months of age via HAZ score and
2. no adequate response despite one month of supplemental feeding, and
3. if there is history of GI illness like chronic or recurrent diarrhea

Exclusion Criteria:

1. no parental consent
2. no anesthesia clearance

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children 6- 24 months
Sampling Method: Probability Sample
Enrollment: 380 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Correlation of Intestinal biomarkers with growth faltering from birth to 24 months | 24 months
  Investigators aimed to validate putative biomarkers of growth faltering, selected based on their role in gut inflammation [fecal myeloperoxidase (MPO) and neopterin (NEO)], enterocyte regeneration (Reg-1b) and proliferation [Glucagon Like Peptide-2 (GLP2)].
Correlation of systemic inflammation biomarkers with growth faltering from birth to 24 months | 24 months
  We also measured the association of a few systemic inflammatory biomarkers [serum Ferritin, c-reactive protein (CRP), α1 acid glycoprotein (AGP)] as well as Insulin-Like Growth factor 1 (IGF-1) with linear growth

CONTACTS AND LOCATIONS:
Overall Officials: Syed Asad Ali, Principal Investigator — Aga Khan University
Locations (1):
- Matiari, Matiari, Sindh, Pakistan